CLINICAL TRIAL: NCT03240406
Title: Multicultural Healthy Diet to Reduce Cognitive Decline & Alzheimer's Disease Risk
Brief Title: Multicultural Healthy Diet to Reduce Cognitive Decline
Acronym: MHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Penn State University (Other); Kaiser Permanente (Other); University of Minnesota (Other); National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Yasmin Mossavar-Rahmani, Professor of Epidemiology & Population Health, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-6613; R01AG055527 (NIH); K99AG056670 (NIH); UL1TR002556 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Diet Modification; Cognitive Decline; Cognitive Change
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Self Care

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized clinical trial to the effects of an anti-inflammatory diet on cognition in a middle-aged cohort. The comparison arm will receive information on self-care matters such as aches and pains of aging.
Who Masked: Outcomes Assessor
Masking Description: The research clinician who assesses cognitive status needs to be blinded to assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory dietary intervention (Active Comparator): 18 month intervention of dietary counseling to adhere to the Multicultural Healthy Diet or the anti-inflammatory diet,
  Interventions: Other: Multicultural Healthy Diet
- Usual Diet plus Self-Care (Placebo Comparator): 18 month intervention of usual diet plus self-care modules
  Interventions: Other: Usual Diet plus Self-Care

INTERVENTIONS:
Other: Multicultural Healthy Diet — An anti-inflammatory dietary pattern consists of a dietary pattern that has high anti-inflammatory potential
  Arms: Anti-inflammatory dietary intervention
Other: Usual Diet plus Self-Care — Usual diet plus sessions that focus on self-care such as dealing with aches and pains of aging.
  Arms: Usual Diet plus Self-Care

SUMMARY:
This is a pilot randomized controlled clinical trial is designed to investigate whether the Multicultural Healthy Diet (MHD), an anti-Inflammatory diet tailored to a multi-cultural population, can improve cognitive functioning in a middle aged (40-65 yr) urban population in Bronx, New York compared to a usual diet.

DETAILED DESCRIPTION:
The Multicultural Healthy Diet (MHD) is a pilot randomized controlled clinical trial designed to test the effects of an 18 month intervention on cognitive function among 290 middle-aged individuals (40-65 yr). MHD is an anti-inflammatory diet tailored to a multicultural population. The emphasis of the intervention is on plant-based foods and limited animal and high saturated fat foods with focus on anti-inflammatory foods/food components specific to the cultural context of the participants. The trial will employ a parallel group design comparing the effects of the dietary intervention (MHD) on cognitive status to those of the control diet or usual diet plus modules on self-care matters such as dealing with aches and pains of aging, obtaining a health care proxy ,etc. To show that MHD can be adapted to this population serum biomarkers indicative of the MHD diet pattern such as fatty acid profile as well as other key nutrition biomarkers will be evaluated. Other aims include testing whether the MHD intervention can benefit cognitive function using real-time ambulatory assessments. The investigators will also assess plasma and serum markers of inflammation. Components of the MHD diet that are associated with stable or improved measures of cognition will also be evaluated. The clinical site for the proposed study is at the Albert Einstein College of Medicine; the ambulatory cognitive assessment reading center is at Pennsylvania State University, State College; the statistical core is at the Kaiser Permanente Washington Health Research Institute and the laboratory for biospecimen analysis is at the University of Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* living, working, attending school or visiting Co-op City, Bronx (e.g. for shopping, doctors' visits, etc.) or communities neighboring Co-op City and between 40-65 yr of age
* willingness to accept assignment to intervention or comparison diet group
* willingness to participate in a study where weight loss is not a primary goal

Exclusion Criteria:

* cognitively impaired
* history of traumatic brain injury
* psychiatric illness
* history of diabetes and experiencing hypoglycemia
* liver disease
* uncontrolled hypertension as defined as blood pressure > 140/90 mm Hg
* history of cardiovascular disease that affects physical functioning
* severe chronic illness
* low literacy
* history of alcohol or drug dependence
* hematologic disease or malignancy not in remission for more than 5 years
* visual, auditory, or motor impairment that precludes cognitive testing.
* chronic kidney disease on dialysis or special diet

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Mossavar-Rahmani, Ph.D, RD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and specimens will be shared with potential collaborators, after obtaining participant consent, consistent with HIPPA guidelines
Supporting Information: Study Protocol
Time Frame: Reasonable time after completion of data analysis and key manuscripts
Access Criteria: Data and specimens will be shared with potential collaborators, after obtaining participant consent, consistent with HIPPA guidelines.

REFERENCES:
- [Background] Mossavar-Rahmani Y, Shaw PA, Hakun JG, Katz MJ, Wylie-Rosett J, Sliwinski MJ. Multicultural Healthy Diet to Reduce Cognitive Decline & Alzheimer's Disease Risk: Study protocol for a pilot randomized controlled trial. Contemp Clin Trials. 2023 Jan;124:107006. doi: 10.1016/j.cct.2022.107006. Epub 2022 Nov 14. PMID 36396064
- [Derived] Mossavar-Rahmani Y, Hyun N, Hakun JG, Katz MJ, Pavlovic JM, Zetterberg H, Wang Z, Yang JB, Wylie-Rosett J, Hebert JR, Sliwinski MJ, Shaw PA. The effects of the Multicultural Healthy Diet on cognitive decline and Alzheimer's disease risk: a phase II randomized controlled trial in middle-aged adults. Am J Clin Nutr. 2025 Jul;122(1):48-59. doi: 10.1016/j.ajcnut.2025.05.011. Epub 2025 May 22. PMID 40412481
- [Derived] Hakun JG, Benson L, Qiu T, Elbich DB, Katz M, Shaw PA, Sliwinski MJ, Mossavar-Rahmani Y. Cognitive Health Benefits of Everyday Physical Activity in a Diverse Sample of Middle-Aged Adults. Ann Behav Med. 2025 Jan 4;59(1):kaae059. doi: 10.1093/abm/kaae059. PMID 39427230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the Covid-19 pandemic, collection of biospecimens and anthropometry data in-person was halted from 3/12/2020 to 7/16/2020; screening visits were administered via Zoom instead of in-person. Group and telephone sessions related to intervention and comparison activities continued via Zoom and telephone during this hiatus and until the end of the study. Recruitment slowed during the pandemic and follow-up was extended to allow all participants to meet their primary endpoint milestone
Pre-assignment Details: Of 393 enrolled patients, 290 met eligibility criteria for randomization and were randomized into the study.
  For this study, Burst time intervals are as follows: Baseline (Burst 1), 9 months (Burst 2), 18 months (Burst 3), and 27 months (Burst 4) post-baseline
  Completion of this study was defined as the first of the following: the completion of all activities through:
  1. Burst 4 (27 months post-baseline) OR
  2. August 30, 2023.
Groups:
- Anti-inflammatory Dietary Intervention (MHD Arm): 18 month intervention of dietary counseling to adhere to the Multicultural Healthy Diet or the anti-inflammatory diet,
  Multicultural Healthy Diet: An anti-inflammatory dietary pattern consists of a dietary pattern that has high anti-inflammatory potential
- Usual Diet Plus Self-Care (Comparison Arm): 18 month intervention of usual diet plus self-care modules
  Usual Diet plus Self-Care: Usual diet plus sessions that focus on self-care such as dealing with aches and pains of aging.
Period: Burst 1 (Baseline)
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Started | 144 | 146
Completed | 144 | 146
Not Completed | 0 | 0
Period: Burst 2 (9 Months)
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Started | 144 | 146
Completed | 126 | 129
Not Completed | 18 | 17
Period: Burst 3 (18 Months)
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Started | 122 (Based on the timing of randomization some participants were not eligible to complete Burst 3 and Burst 4.) | 126 (Based on the timing of randomization some participants were not eligible to complete Burst 3 and Burst 4.)
Completed | 98 | 93
Not Completed | 24 | 33
Period: Burst 4 (27 Months)
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Started | 77 (Based on the timing of randomization some participants were not eligible to complete Burst 3 and Burst 4.) | 72 (Based on the timing of randomization some participants were not eligible to complete Burst 3 and Burst 4.)
Completed | 57 | 57
Not Completed | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm) | Total
Number analyzed (Participants) | 144 | 146 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (7.2) | 54.0 (7.0) | 53.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 115 | 230
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 58 | 118
  Not Hispanic or Latino | 84 | 88 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 63 | 67 | 130
  White | 34 | 32 | 66
  More than one race | 28 | 33 | 61
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 144 | 146 | 290

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Global Composite Cognition Score From Baseline
Description: Change in global composite cognition score (standardized unit) is computed as the average of the three domain-specific Z-scores of the participant's performance on three ambulatory cognitive assessments: visuospatial working memory (Dot Grid Memory), processing speed (Symbol Search), and short-term associative memory binding (Color Shapes Task) at 9 months post baseline (Burst 1). Z-scores are centered at a population mean of "0" (i.e., a Z-score of "0" signifies that the data point(s) is equal to the population mean at study baseline for all three tasks in the composite average; positive Z-score group values indicate the number of standard deviations the data point(s) is above the mean and negative Z-score group values indicate the number of standard deviations the data point(s) is below the mean). Mean change in global composite Z-score from baseline will be reported by study arm. Increase in composite Z-scores from baseline are associated with improved cognition.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Participants completing at least 18 sessions for the primary three domains at Bursts 1 or 2 were analyzed. Missing and non-compliant data were multiply imputed using multivariate imputation by chained equations (MICE).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
Z-score | 0.2 (0.8) | 0.2 (0.8)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.259, ANCOVA — Test of the between arm difference in the global composite at Burst 2, adjusted for the study arm, baseline (Burst 1) global composite, and the randomization stratification factors (baseline sex, age, and years of education); ANCOVA of Burst 2 composite adjusted for arm, Burst 1 composite, sex, age, and education. Missing/invalid data were multiply imputed using MICE; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.15 to 0.04] — Mean Difference of MHD Arm compared to control

2. Secondary Outcome: Dietary Inflammatory Index (DII) Score
Description: DII score was determined by an algorithm that summarized the inflammatory potential of the diet. The DII score represents a weighted sum of the self-reported quantities of 28 foods, each translated into Z-scores using a global comparative database consisting of data from 11 countries by subtracting from the individual's self-report value the mean of the global database, then dividing by the standard deviation (SD). Z-scores are centered at a population mean of "0" (i.e., a Z-score of "0" signifies that the data point(s) is = to the population mean at study baseline for all 3 tasks in the composite average; positive and negative Z-score group values indicate the number of SD the data point(s) is above or below the mean, respectively). For this study, possible scoring range for 28 food parameters was -8 to 8 based on ref: Hebert JR, et.al., Perspective: The Dietary Inflammatory Index (DII®): Adv Nutr. 2019;10:185-95. Higher Z-score values are indicative of a more pro-inflammatory diet.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1 (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
Z-score
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 1.10 (1.85) | 1.17 (1.83)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.70 (2.01) | 1.38 (1.76)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.001, ANCOVA — MHD-Comparison difference in Burst 2 value estimated by ANCOVA, adjusted for Burst 1 value, age, sex, years of education; MHD-Comparison difference in Burst 2 value estimated by ANCOVA, adjusted for Burst 1 value, age, sex, years of education; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.02 to -0.27] — Mean Difference of MHD Arm vs Comparison Arm

3. Secondary Outcome: Energy-Adjusted DII Score
Description: Energy-adjusted DII score was determined by an algorithm that summarized the inflammatory potential of the diet. This score represents a weighted sum of self-reported quantities of 28 foods per 1000 kilocalories of consumption that were then translated into Z-scores using a global comparative database of data from 11 countries by subtracting from the individual's self-report value the mean of the global database, then dividing by the SD. Z-scores are centered at a population mean of 0 (i.e., a Z-score of 0 signifies that the data point is = to the population mean at study baseline for all 3 tasks in the composite average; positive and negative Z-score group values indicate the number of SD the data point is above or below the mean, respectively). For this study, possible scoring range for 28 food parameters was -8 to 8 based on ref: Hebert JR, et.al., Perspective: The Dietary Inflammatory Index (DII®): Adv Nutr. 2019;10:185-95. Higher values are indicative of a more inflammatory diet.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1 (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
Z-score
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | -0.30 (1.96) | -0.30 (2.03)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | -0.98 (2.16) | -0.09 (2.03)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p < 0.001, ANCOVA — Estimated from ANCOVA model adjusted for baseline value, age, sex, and years of education at baseline; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.94, 95% CI 2-sided [-1.34 to -0.54] — Mean Difference of MHD Arm vs Comparison Arm

4. Secondary Outcome: Total Serum Folate Levels
Description: Blood sera specimens were collected and processed at Baseline and 9-months post-intervention and shipped to University of Minnesota Advanced Research & Diagnostic Laboratory (ARDL) for total folate analysis by a validated serum folate assay. Mean total folate levels are summarized by study arm and reported in nmol/L. The lower limit of detection (LLOD) for mean total folate is 4.54 nmol/L and the upper limit of detection (ULOD) 90.8 nmol/L. Increase in this biomarker from baseline for MHD participants indicates possible adherence to an MHD dietary pattern such as eating more green leafy vegetables.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: Burst 1, MHD (N=13); Burst 1, Comparison (N=12). Burst 2, MHD (N=36), Burst 2, Comparison (N=44).
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 131 | 134
nmol/L
  Burst 1 (Baseline) | 35.93 (17.19) | 34.72 (15.74)
  Burst 2 (9 months): number analyzed (Participants) | 108 | 102
  Burst 2 (9 months) | 35.26 (17.8) | 35.01 (15.78)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.904, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.24, 95% CI 2-sided [-3.63 to 4.11] — Mean Difference of MHD Arm vs Comparison Arm

5. Secondary Outcome: α-Tocopherol Levels
Description: Blood plasma specimens were collected and processed at Baseline and 9-months post-intervention and shipped to University of Minnesota ARDL for α-tocopherol analysis by an HPLC method. α-Tocopherols were measured with a diode array detector equipped HPLC system. Mean α-tocopherol levels are summarized by study arm and reported in mcg/mL. There are no reference ranges for this biomarker from this laboratory (other than non-negative values). Increase in this biomarker from baseline for MHD participants indicates possible adherence to an MHD dietary pattern.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: Burst 1, MHD (N=7); Burst 1, Comparison (N=6). Burst 2, MHD (N=31), Burst 2, Comparison (N=38).
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 137 | 140
mcg/mL
  Burst 1 (Baseline) | 11.39 (3.49) | 11.02 (2.94)
  Burst 2 (9 Months): number analyzed (Participants) | 113 | 108
  Burst 2 (9 Months) | 11.45 (3.73) | 11.26 (3.56)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.721, ANCOVA — MHD-Comparison difference in Burst 2 value estimated by ANCOVA, adjusted for Burst 1 value, age, sex, and education; tocopherol biomarker values additionally adjusted for Burst 1 and Burst 2 levels of HDL, LDL, and triglycerides; Burst 2 value estimated by ANCOVA, adjusted for Burst 1 value, age, sex, years of education; Burst 1 and Burst 2 levels of HDL, LDL and triglycerides; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.76 to 0.52] — Mean Difference of MHD Arm vs Comparison Arm

6. Secondary Outcome: α-Carotenoid Levels
Description: Blood plasma specimens were collected and processed at Baseline and 9-months post-intervention from a sub-sample and shipped to University of Minnesota ARDL lab for α-carotenoid analysis by an HPLC method. α-Carotenoids were measured with a diode array detector equipped HPLC system. Mean α-carotenoid levels are summarized by study arm and reported in mcg/mL. There are no reference ranges for this biomarker (other than non-negative values). Increase in this biomarker from baseline for MHD participants indicates possible adherence to an MHD dietary pattern.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: Burst 1, MHD (N=7); Burst 1, Comparison (N=6). Burst 2, MHD (N=31), Burst 2, Comparison (N=38).
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 137 | 140
mcg/mL
  Burst 1 (Baseline) | 0.04 (0.04) | 0.04 (0.03)
  Burst 2 (9 Months): number analyzed (Participants) | 113 | 108
  Burst 2 (9 Months) | 0.04 (0.04) | 0.04 (0.06)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.769, ANCOVA — MHD-Comparison difference in Burst 2 value estimated by ANCOVA, adjusted for Burst 1 value, age, sex, and education; carotenoid biomarker values additionally adjusted for Burst 1 and Burst 2 levels of HDL, LDL, and triglycerides; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.01 to 0.01] — Mean Difference of MHD Arm vs Comparison Arm

7. Secondary Outcome: Vitamin B12 Levels
Description: Blood sera specimens were collected and processed at Baseline and 9-months post-intervention and shipped to University of Minnesota ARDL laboratory for Vitamin B12 analysis by a validated Vitamin B12 assay. Mean Vitamin B12 levels are summarized by study arm and reported in pg/mL. Reference ranges for this biomarker are: 232-1245 pg/mL and LLOD is 100 pg/mL. Increase in this biomarker from baseline for MHD participants indicates possible adherence to an MHD dietary pattern.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: Burst 1, MHD (N=10); Burst 1, Comparison (N=7). Burst 2, MHD (N=33), Burst 2, Comparison (N=40).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 134 | 139
pg/mL
  Burst 1 (Baseline) | 736.78 (513.94) | 712.89 (445.71)
  Burst 2 (9 Months): number analyzed (Participants) | 111 | 106
  Burst 2 (9 Months) | 718.23 (522.58) | 716.22 (417.64)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.978, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.37, 95% CI 2-sided [-100.13 to 97.4] — Mean Difference of MHD Arm vs Comparison Arm

8. Secondary Outcome: Fatty Acid Profile
Description: Blood plasma specimens were collected and processed at Baseline and 9-months follow-up for a sub-sample and shipped to University of Minnesota ARDL laboratory for total fatty acid analysis by a gas chromatography method. Fatty acids are expressed as a percent of total fatty acids. Fatty acids are compared with each sample rather than measured against a standard and the range of percentage values for each fatty acid is 0-100%. Mean percentage plasma levels of the following fatty acids will be summarized by study arm for Burst 2: Sum of monounsaturated fatty acids (n=6); Long chain saturated fatty acids (fatty acids with 20 or more carbons (n=3)); EPA (eicosapentaenoic acid); DHA (docosahexaenoic acid); n3 DPA (omega three docosapentaenoic acid).
  Monounsaturated fat is a composite of 6 fatty acids: 16:1n7 cis, 17:1n7T, 18:1n9 cis,18:1n7 cis, 20:1n9, and 24:1n9 Long chain saturated fat is a composite of 3 fatty acids: 22:0, 23:0, and 24:0
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=61); MHD, Burst 2 (N=52). Comparison, Burst 1 (N=61); Comparison, Burst 2 (N=52). For the Fatty Acid Profile Outcome Measure only a subset of samples were analyzed due to cost.
Measure: Mean (Standard Deviation); unit: % of total fatty acid
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 83 | 94
% of total fatty acid
  Monounsaturated Fat at Burst 1 (Baseline) | 10.76 (1.30) | 11.09 (1.67)
  Monounsaturated Fat at Burst 2 (9 Months) | 10.91 (1.44) | 10.96 (1.58)
  Long-chain Saturated Fat at Burst 1 (Baseline) | 2.14 (0.38) | 2.12 (0.45)
  Long-chain Saturated Fat at Burst 2 (9 Months) | 2.15 (0.41) | 2.23 (0.42)
  EPA at Burst 1 (Baseline) | 0.98 (1.24) | 0.90 (0.45)
  EPA at Burst 2 (9 Months) | 1.01 (0.90) | 0.85 (0.44)
  DHA at Burst 1 (Baseline) | 3.67 (1.09) | 3.65 (1.30)
  DHA at Burst 2 (9 Months) | 3.77 (1.41) | 3.48 (1.05)
  n3 DPA at Burst 1 (Baseline) | 1.10 (0.18) | 1.09 (0.21)
  n3 DPA at Burst 2 (9 Months) | 1.07 (0.17) | 1.07 (0.18)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Statistical Analysis results for Monounsaturated Fat; Test type: Superiority; p = 0.395, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.2 to 0.51] — Mean Difference of MHD Arm vs Comparison Arm
Statistical Analysis 2: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Statistical Analysis results for Long Chain Saturated Fat; Test type: Superiority; p = 0.019, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.21 to -0.02] — Mean Difference of MHD Arm vs Comparison Arm
Statistical Analysis 3: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Statistical Analysis results for EPA; Test type: Superiority; p = 0.201, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.07 to 0.31] — Mean Difference of MHD Arm vs Comparison Arm
Statistical Analysis 4: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Statistical Analysis results for DHA; Test type: Superiority; p = 0.039, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.27, 95% CI 2-sided [0.01 to 0.53] — Mean Difference of MHD Arm vs Comparison Arm
Statistical Analysis 5: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Statistical Analysis results for n3 DPA; Test type: Superiority; p = 0.619, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.06 to 0.03] — Mean difference of MHD Arm vs Comparison Arm

9. Secondary Outcome: Serum Sodium
Description: Serum specimens were collected and processed at Baseline and 9-months follow-up and shipped to University of Minnesota ARDL laboratory for analysis on Roche Cobas 8000 Chemistry Analyzer. Mean serum sodium levels are summarized by study arm and reported in mmol/L. Reference range is 136-145 mmol/L and the lower LOD is 80 mmol/L. Decreased serum sodium levels from baseline may indicate dehydration.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: Burst 1, MHD: (N=10); Burst 1, Comparison: (N=7). Burst 2, MHD: (N=33); Burst 2, Comparison: (N=40)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 134 | 139
mmol/L
  Burst 1 (Baseline) | 139.88 (1.88) | 139.89 (1.91)
  Burst 2 (9 Months): number analyzed (Participants) | 111 | 106
  Burst 2 (9 Months) | 140.24 (2.4) | 140.11 (1.99)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.521, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.18, 95% CI 2-sided [-0.37 to 0.73] — Mean Difference of MHD Arm vs Comparison Arm

10. Secondary Outcome: Self-reported Diet Components and Food Groups: Total Moisture
Description: Total Moisture obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Total moisture from diet was captured by the MOIS variable field within the ASA24. This field is quantified in grams (g) of water. Possible results values are limited to values > 0 (i.e., positive values). Basic descriptive statistics were used to summarize data by arm.ASA-2018 and 2020
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 1821 (840) | 1812 (791)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 1943 (959) | 1790 (815)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.101, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 145.0, 95% CI 2-sided [-27.7 to 317.6] — Mean Difference of MHD Arm vs Comparison Arm

11. Secondary Outcome: Self-reported Diet Components and Food Groups: Energy
Description: Energy obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Total energy from diet was captured by the KCAL variable field within the ASA24. This field represents kilocalories (kcal) of energy. Possible results values are to values > 500kcal. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1 (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2, (N=22).
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
kcal
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 1622.31 (574.26) | 1608.62 (518)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 1545.25 (552.32) | 1560.3 (532.73)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.645, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -24.63, 95% CI 2-sided [-129.16 to 79.89] — Mean Difference of MHD Arm vs Comparison Arm

12. Secondary Outcome: Self-reported Diet Components and Food Groups: Protein
Description: Protein obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Protein from the diet was captured by the PROT variable field within the ASA24. This field represents grams (g) of protein consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1 (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2, (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 73.92 (27.21) | 73.31 (23.62)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 73.42 (24.5) | 70.09 (27.31)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.245, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 3.26, 95% CI 2-sided [-2.23 to 8.75] — Mean Difference of MHD Arm vs Comparison Arm

13. Secondary Outcome: Self-reported Diet Components and Food Groups: Total Intact Fruits + Fruit Juices
Description: Total Intact fruits and fruit juices obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Total Intact fruit and fruit juice consumption from the diet was captured by the F_TOTAL variable field within the ASA24. This field represents total fruit consumption in cup equivalents (cup eq). Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: cup eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
cup eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.85 (0.91) | 0.77 (0.78)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.95 (0.92) | 0.68 (0.76)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.032, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.21, 95% CI 2-sided [0.02 to 0.4] — Mean Difference of MHD Arm vs Comparison Arm

14. Secondary Outcome: Self-reported Diet Components and Food Groups: Dark Green Vegetables
Description: Dark Green Vegetables obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Dark green vegetable consumption from the diet was captured by the V_DRKGR variable field within the ASA24. This field represents dark green vegetable consumption in cup equivalents (cup eq). Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: cup eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
cup eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.3 (0.33) | 0.33 (0.34)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.43 (0.45) | 0.28 (0.28)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.17, 95% CI 2-sided [0.08 to 0.26] — Mean Difference of MHD Arm vs Comparison Arm

15. Secondary Outcome: Self-reported Diet Components and Food Groups: Total Fats
Description: Total fats obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Total fats from the diet, which consisted of total saturated fatty acids, total monounsaturated fatty acids, and total polyunsaturated fatty acids, was captured by the TFAT variable field within the ASA24. This field represents grams (g) of total fats consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 67.3 (26.52) | 66.71 (25.45)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 65.69 (29.13) | 66.77 (25.4)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.635, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.36, 95% CI 2-sided [-6.95 to 4.24] — Mean Difference of MHD Arm vs Comparison Arm

16. Secondary Outcome: Self-reported Diet Components and Food Groups: Solid Fats
Description: Solid fats obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Solid fats from the diet was captured by the DISCFAT_SOL variable field within the ASA24. This field represents grams (g) of solid fats consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 26.84 (15.44) | 26.77 (14.68)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 23.14 (15.44) | 26.93 (14.48)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.019, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -3.52, 95% CI 2-sided [-6.44 to 0.59] — Mean Difference of MHD Arm vs Comparison Arm

17. Secondary Outcome: Self-reported Diet Components and Food Groups: Carbohydrates
Description: Carbohydrates obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Carbohydrates from the diet was captured by the CARB variable field within the ASA24. This field represents grams (g) of carbohydrates consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 2 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 2 (Baseline) | 181.11 (74.37) | 176.49 (66.03)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 169.66 (71.27) | 169.23 (67.2)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.639, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -3.13, 95% CI 2-sided [-16.18 to 9.92] — Mean Difference of MHD Arm vs Comparison Arm

18. Secondary Outcome: Self-reported Diet Components and Food Groups: Total Folate From Food
Description: Total Folate from food obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Total Folate from food was captured by the FF variable field within the ASA24. This field represents micrograms (mcg) of total folate from food consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 199.05 (93.83) | 197.56 (93.23)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 224.17 (110.14) | 181.69 (83.24)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 41.71, 95% CI 2-sided [21.47 to 61.96] — Mean Difference of MHD Arm vs Comparison Arm

19. Secondary Outcome: Self-reported Diet Components and Food Groups: Non-food Folate
Description: Non-food Folate obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Non-food Folate was captured by the FDFE variable field within the ASA24. This field represents micrograms (mcg) of Non-food Folate consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 125.15 (86.02) | 130.78 (108.64)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 109.97 (80.89) | 127.73 (98.76)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.115, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -15.37, 95% CI 2-sided [-34.44 to 3.69] — Mean Difference of MHD Arm vs Comparison Arm

20. Secondary Outcome: Self-reported Diet Components and Food Groups: Vitamin B-12
Description: Vitamin B-12 obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Vitamin B-12 was captured by the VB12 variable field within the ASA24. This field represents micrograms (mcg) of Vitamin B-12 consumed (including supplemental sources). Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 4.25 (2.59) | 4.21 (2.64)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 4.18 (2.63) | 4.06 (2.43)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.847, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.53 to 0.64] — Mean Difference of MHD Arm vs Comparison Arm

21. Secondary Outcome: Self-reported Diet Components and Food Groups: Alpha Carotene
Description: Alpha Carotene obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Alpha Carotene from the diet was captured by the ACAR variable field within the ASA24. This field represents micrograms (mcg) of Alpha Carotene consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 568.66 (900.88) | 448.66 (676.44)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 586.56 (858.46) | 392.19 (626.37)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.191, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 118.57, 95% CI 2-sided [-58.62 to 295.76] — Mean Difference of MHD Arm vs Comparison Arm

22. Secondary Outcome: Self-reported Diet Components and Food Groups: Beta Carotene
Description: Beta Carotene obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Beta Carotene from the diet was captured by the BCAR variable field within the ASA24. This field represents micrograms (mcg) of Beta Carotene consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 3464.67 (3758.65) | 3389.68 (4072.72)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 4040.06 (3887.57) | 2948.25 (2823.76)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.019, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 955.19, 95% CI 2-sided [164.63 to 1745.74] — Mean Difference of MHD Arm vs Comparison Arm

23. Secondary Outcome: Self-reported Diet Components and Food Groups: Retinol
Description: Retinol obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Retinol from the diet was captured by the RET variable field within the ASA24. This field represents micrograms (mcg) of Retinol consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 327.45 (210.72) | 317.48 (190.29)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 302.99 (181.71) | 318.97 (210.58)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.493, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -15.74, 95% CI 2-sided [-60.66 to 29.19] — Mean Difference of MHD Arm vs Comparison Arm

24. Secondary Outcome: Self-reported Diet Components and Food Groups: Beta Cryptoxanthin
Description: Beta Cryptoxanthin obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Beta Cryptoxanthin from the diet was captured by the CRYP variable field within the ASA24. This field represents micrograms (mcg) of Beta Cryptoxanthin consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 96.49 (166.36) | 57.57 (84.37)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 81.28 (111.66) | 57.41 (63.53)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.18, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 14.83, 95% CI 2-sided [-6.78 to 36.45] — Mean Difference of MHD Arm vs Comparison Arm

25. Secondary Outcome: Self-reported Diet Components and Food Groups: Lycopene
Description: Lycopene obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Lycopene from the diet was captured by the LYCO variable field within the ASA24. This field represents micrograms (mcg) of Lycopene consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 3905.68 (5106.71) | 3558.21 (3819.37)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 3685.28 (4671.61) | 3244.35 (2902.16)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.379, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 436.14, 95% CI 2-sided [-534.05 to 1406.33] — Mean Difference of MHD Arm vs Comparison Arm

26. Secondary Outcome: Self-reported Diet Components and Food Groups: Lutein + Zeaxanthin
Description: Lutein + Zeaxanthin obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Lutein + Zeaxanthin from the diet was captured by the LZ variable field within the ASA24. This field represents micrograms (mcg) of Lutein + Zeaxanthin consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mcg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 2885.48 (3661.72) | 2765.1 (4110.87)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 3570.56 (4028.1) | 2609.09 (3357.6)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.083, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 784.06, 95% CI 2-sided [-99.73 to 1667.85] — Mean Difference of MHD Arm vs Comparison Arm

27. Secondary Outcome: Self-reported Diet Components and Food Groups: Alpha Tocopherol (Vitamin E)
Description: Alpha Tocopherol (Vitamin E) obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Alpha Tocopherol from the diet was captured by the ATOC variable field within the ASA24. This field represents micrograms (mg) of Alpha Tocopherol consumed (including from supplemental sources). Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
mg
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 7.48 (3.07) | 7.59 (3.87)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 8.69 (5.34) | 7.34 (3.41)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.011, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 1.33, 95% CI 2-sided [0.32 to 2.35] — Mean Difference of MHD Arm vs Comparison Arm

28. Secondary Outcome: Self-reported Diet Components and Food Groups: Seafood High in n-3 Fatty Acids
Description: Seafood high in n-3 fatty acids obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Seafood high in n-3 fatty acids from the diet was captured by the M_FISH_HI variable field within the ASA24. This field represents ounce equivalents (oz eq) of Seafood high in n-3 fatty acids consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: oz eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
oz eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.58 (0.94) | 0.44 (0.92)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.56 (1.06) | 0.44 (0.9)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.541, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.16 to 0.31] — Mean Difference of MHD Arm vs Comparison Arm

29. Secondary Outcome: Self-reported Diet Components and Food Groups: EPA (P205)
Description: EPA (P205) obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. EPA (P205) from the diet was captured by the P205 variable field within the ASA24. This field represents grams (g) of EPA (P205) consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.07 (0.01) | 0.06 (0.08)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.07 (0.08) | 0.05 (0.07)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.273, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.01 to 0.03] — Mean Difference of MHD Arm vs Comparison Arm

30. Secondary Outcome: Self-reported Diet Components and Food Groups: DHA (P226)
Description: DHA (P226) obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. DHA (P226) from the diet was captured by the P226 variable field within the ASA24. This field represents grams (g) of DHA (P226) consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.14 (0.17) | 0.12 (0.16)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.13 (0.16) | 0.1 (0.12)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.116, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.01 to 0.06] — Mean Difference of MHD Arm vs Comparison Arm

31. Secondary Outcome: Self-reported Diet Components and Food Groups: DPA (P225)
Description: DPA (P225) obtained from the participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. DPA (P225) from the diet was captured by the P225 variable field within the ASA24. This field represents grams (g) of DPA (P225) consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
g
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.03 (0.03) | 0.03 (0.03)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.03 (0.03) | 0.02 (0.02)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.213, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0.01] — Mean Difference of MHD Arm vs Comparison Arm

32. Secondary Outcome: Self-reported Diet Components and Food Groups: Beans and Peas (Legumes)
Description: Beans and peas (Legumes) consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Legumes information from the diet was captured by the V_LEGUMES variable field within the ASA24. This field represents cup equivalents (cup eq) of legumes consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: cup eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
cup eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.12 (0.17) | 0.1 (0.16)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.14 (0.22) | 0.09 (0.14)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.036, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [0 to 0.09] — Mean Difference of MHD Arm vs Comparison Arm

33. Secondary Outcome: Self-reported Diet Components and Food Groups: Whole Grains
Description: Whole grains consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Whole grains information from the diet was captured by the G_WHOLE variable field within the ASA24. This field represents ounce equivalents (oz eq) of whole grains consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: oz eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
oz eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.75 (0.76) | 0.85 (0.93)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 1.06 (1.17) | 0.90 (1.01)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.223, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.1 to 0.43] — Mean Difference of MHD Arm vs Comparison Arm

34. Secondary Outcome: Self-reported Diet Components and Food Groups: Cured Meats
Description: Cured meats consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Cured meats information from the diet was captured by the PF_CUREDMEAT variable field within the ASA24. This field represents ounce equivalents (oz eq) of cured meats consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: oz eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
oz eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.74 (0.93) | 0.64 (0.83)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.63 (0.82) | 0.76 (0.95)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.119, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.38 to 0.04] — Mean Difference of MHD Arm vs Comparison Arm

35. Secondary Outcome: Self-reported Diet Components and Food Groups: Poultry
Description: Poultry consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Poultry information from the diet was captured by the PF_POULT variable field within the ASA24. This field represents ounce equivalents (oz eq) of poultry consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: oz eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
oz eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 1.82 (1.65) | 1.89 (1.64)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 1.79 (1.56) | 1.82 (1.54)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.841, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.41 to 0.33] — Mean Difference of MHD Arm vs Comparison Arm

36. Secondary Outcome: Self-reported Diet Components and Food Groups: Nuts and Seeds
Description: Nuts and seeds consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Nuts and seeds information from the diet was captured by the PF_NUTSDS variable field within the ASA24. This field represents ounce equivalents (oz eq) of nuts and seeds consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: oz eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
oz eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.57 (0.91) | 0.58 (0.94)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.82 (1.43) | 0.56 (0.88)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.088, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.04 to 0.53] — Mean Difference of MHD Arm vs Comparison Arm

37. Secondary Outcome: Self-reported Diet Components and Food Groups: Cheeses
Description: Cheeses consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Cheese information from the diet was captured by the D_CHEESE variable field within the ASA24. This field represents cup equivalents (cup eq) of cheeses consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: cup eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
cup eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 0.58 (0.48) | 0.62 (0.6)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 0.51 (0.54) | 0.54 (0.48)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.893, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.13 to 0.11] — Mean Difference of MHD Arm vs Comparison Arm

38. Secondary Outcome: Self-reported Diet Components and Food Groups: Added Sugars
Description: Added sugars consumed as part of participants' diet was derived as a parameter of the self-reported diet components and food groups from the 2018 and 2020 versions of the Automated Self-reported Self-administered 24 hour food records (ASA24-2018 and ASA24-2020) at baseline and 9 month follow-up. Added sugars information from the diet was captured by the ADD_SUGARS variable field within the ASA24. This field represents tablespoon equivalents (tsp eq) of added sugars consumed. Possible results values are limited to non-negative values. Basic descriptive statistics were used to summarize data by arm.
Time Frame: Baseline (Burst 1) and 9 months (Burst 2)
Population: Missing data: MHD, Burst 1, (N=1); MHD, Burst 2 (N=19). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=22).
Measure: Mean (Standard Deviation); unit: tsp eq
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 144 | 146
tsp eq
  Burst 1 (Baseline): number analyzed (Participants) | 143 | 146
  Burst 1 (Baseline) | 10.06 (7.57) | 9.91 (6.79)
  Burst 2 (9 Months): number analyzed (Participants) | 125 | 124
  Burst 2 (9 Months) | 7.91 (6.02) | 9.31 (6.89)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.042, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.43, 95% CI 2-sided [-2.81 to -0.06] — Mean Difference of MHD Arm vs Comparison Arm

39. Secondary Outcome: Symbol Search Task Performance
Description: Symbol Search Task Performance is an ambulatory cognitive assessment of processing speed/attention. The task is administered 5 times daily throughout each 7-day measurement Burst (Baseline, 9 months, 18 months, 27 months). Mean response time in milliseconds (ms) for accurate trials will be determined and reported. Possible values ranges for Symbol Search Task Performance are >0 ms (i.e., positive values). Lower Symbol Search Task Performance values in mean response time are indicative of improvement in cognitive processing.
Time Frame: Baseline (Burst 1), and 9 months (Burst 2), 18 months (Burst 3), and 27 months (Burst 4) post-intervention
Population: Missing data: MHD, Burst 1, (N=4); MHD, Burst 2 (N=29); MHD, Burst 3 (N=24); MHD, Burst 4 (N=20). Comparison, Burst 1 (N=0); Comparison, Burst 2 (N=31); Comparison, Burst 3 (N=34); Comparison, Burst 4 (N=15).
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 140 | 146
ms
  Burst 1 (Baseline) | 1,874.7 (474.3) | 1,846.4 (466.3)
  Burst 2 (9 months): number analyzed (Participants) | 115 | 115
  Burst 2 (9 months) | 1,854.4 (537.5) | 1,800.5 (457.8)
  Burst 3 (18 months): number analyzed (Participants) | 98 | 92
  Burst 3 (18 months) | 1,845.0 (465.6) | 1,825.6 (470.7)
  Burst 4 (27 months): number analyzed (Participants) | 57 | 57
  Burst 4 (27 months) | 1,765.2 (529.3) | 1,812.0 (445.0)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.031, Mixed Models Analysis — Linear mixed-effects model adjusted for adjusted for arm, year, weekday, season, EMA cognition, baseline age, sex, education yrs, # of sessions (cubic spline), and time of day (cubic spline); Adjusted for arm, year, weekday, season, EMA cognition, baseline age, sex, education yrs, # of sessions (cubic spline), and time of day (cubic spline); Slope = -16, 95% CI 2-sided [-31 to -1.5] — Difference in the slopes of processing speed over years between MHD Arm and Comparison Arm

40. Secondary Outcome: Grid Memory Task Performance
Description: Grid Memory Task Performance is an ambulatory cognitive assessment of visuospatial working memory. The task is administered 5 times daily throughout each 7-day measurement Burst (Baseline, 9 months, 18 months, 27 months). The mean error distance (pixel Euclidean distance, represented in pixels) of the red dots between study and recall arrays will be quantified and reported based on the completion of 4 trials. Possible value ranges for pixels are >0 (i.e., positive values). Lower pixel values are indicative of improved short-term recall and visuospatial working memory.
Time Frame: Baseline (Burst 1), and 9 months (Burst 2), 18 months (Burst 3), and 27 months (Burst 4) post-intervention
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 140 | 146
pixels
  Burst 1 (Baseline) | 34.0 (15.6) | 35.2 (15.3)
  Burst 2 (9 months): number analyzed (Participants) | 115 | 115
  Burst 2 (9 months) | 29.0 (14.7) | 30.4 (15.4)
  Burst 3 (18 months): number analyzed (Participants) | 98 | 92
  Burst 3 (18 months) | 26.8 (15.5) | 31.6 (15.8)
  Burst 4 (27 months): number analyzed (Participants) | 57 | 57
  Burst 4 (27 months) | 25.6 (15.7) | 27.4 (16.3)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.55, Mixed Models Analysis — Linear mixed-effects model adjusted for arm, year, weekday, season, EMA cognition, baseline age, sex, education yrs, # of sessions (cubic spline), and time of day (cubic spline); [statistical method as in outcome 39, analysis 1]; Slope = 0.12, 95% CI 2-sided [-0.27 to 0.51] — Difference in the slopes of error distance over years between MHD Arm vs Comparison Arm

41. Secondary Outcome: Color Shapes Task Performance
Description: Color Shapes Task Performance is an ambulatory cognitive assessment of short-term associative visual memory. The task is administered 5 times daily throughout each 7-day measurement Burst. The task had 2 conditions, signal present and signal absent. Hit rate represents the proportion of trials where participants correctly responded that signal was present. False alarm rate represents the proportion of trials where a signal was absent where participants incorrectly responded that a signal was present. Corrected Recognition Score represents the overall sensitivity to the signal and is calculated by subtracting the False alarm rate from the Hit rate and is summarized by study arm as described in Hakun, et.al., (2024). Mobile Monitoring of Cognitive Change (M2C2): High-Frequency Assessments and Protocol Reporting Guidelines. Possible ranges for Corrected Recognition Score are -1 to 1. Higher Corrected Recognition Rate values are indicative of better short term associative memory-binding.
Time Frame: Baseline (Burst 1), and 9 months (Burst 2), 18 months (Burst 3), and 27 months (Burst 4) post-intervention
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Corrected Recognition Score
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
Number analyzed (Participants) | 140 | 146
Corrected Recognition Score
  Burst 1 (Baseline) | 0.6 (0.2) | 0.6 (0.2)
  Burst 2 (9 months): number analyzed (Participants) | 115 | 115
  Burst 2 (9 months) | 0.6 (0.2) | 0.6 (0.2)
  Burst 3 (18 months): number analyzed (Participants) | 98 | 92
  Burst 3 (18 months) | 0.6 (0.2) | 0.6 (0.2)
  Burst 4 (27 months): number analyzed (Participants) | 57 | 57
  Burst 4 (27 months) | 0.7 (0.2) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Anti-inflammatory Dietary Intervention (MHD Arm) vs Usual Diet Plus Self-Care (Comparison Arm); Test type: Superiority; p = 0.846, Generalized Estimating Equation — Generalized Estimating equation Poisson model adjusted for arm, year, weekday vs weekend, season, EMA cognition, baseline age, sex, education yrs, # of sessions (cubic spline), time of day (cubic spline); Adjusted for arm, year, wkday/wknd, season, EMA cognition, baseline age, sex, education yrs, # of sessions (cubic spline), time of day (cubic spline); Slope = -0.018, 95% CI 2-sided [-0.090 to 0.054] — Difference in the slopes of log-transformed error rates over years between the MHD Arm and the Comparison Arm

ADVERSE EVENTS:
Time Frame: Adverse event data was collected every 9 months, up to 27 months total
Arm/Group | Anti-inflammatory Dietary Intervention (MHD Arm) | Usual Diet Plus Self-Care (Comparison Arm)
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/146
Serious Adverse Events (participants affected / at risk) | 9/144 | 10/146
Other Adverse Events (participants affected / at risk) | 73/144 | 71/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-inflammatory Dietary Intervention (MHD Arm) (N=144) | Usual Diet Plus Self-Care (Comparison Arm) (N=146)
Hospitalization for COVID-19 (Infections and infestations) | 1 | 4 — Verbatim Term
Breast Cancer, Surgery and Chemotherapy (Surgical and medical procedures) | 0 | 4 — Verbatim Term
Hospitalization for Stress (Nervous system disorders) | 0 | 1 — Verbatim Term
Treatment for Brain Cancer (Surgical and medical procedures) | 0 | 1 — s/p Brain tumor surgery prior to enrollment
Hospitalization for Stent Placement (Surgical and medical procedures) | 1 | 0 — Verbatim Terms
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Verbatim Term(s)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Verbatim Term(s)
Pancreatitis (Gastrointestinal disorders) | 1 | 0 — Verbatim Term
Congestive Heart Failure (Cardiac disorders) | 1 | 0 — Verbatim Term(s)
Acute Renal Failure (Renal and urinary disorders) | 1 | 0 — s/p Chronic Kidney Disease
Heart Attack, Heart Surgery (Cardiac disorders) | 1 | 0 — Verbatim Terms
Gastric Bypass Revision (Surgical and medical procedures) | 1 | 0 — Verbatim Term(s)
Emergent Visit for Gastric Bypass (Surgical and medical procedures) | 1 | 0 — Verbatim Term(s). s/p Gastric Bypass Surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-inflammatory Dietary Intervention (MHD Arm) (N=144) | Usual Diet Plus Self-Care (Comparison Arm) (N=146)
Respiratory Problems (Respiratory, thoracic and mediastinal disorders) | 2 | 2 — Verbatim Term(s)
Headache (Nervous system disorders) | 8 | 8
High Blood Pressure (Vascular disorders) | 20 | 18 — Verbatim Term(s)
Periodontal Disease (Gastrointestinal disorders) | 3 | 1
Osteoarthritis, Fibromyalgia/Osteoarthritis, muscular or bone problems (Musculoskeletal and connective tissue disorders) | 10 | 8 — Verbatim Terms
Obesity (Metabolism and nutrition disorders) | 1 | 0
Stomach or Bowel Issues (Gastrointestinal disorders) | 3 | 7 — Verbatim Terms
Hearing or Vision Problems (Ear and labyrinth disorders) | 15 | 17 — Verbatim Terms. Includes Ear and Eye Disorders
Blood Circulation or Blood-Related Problems (Blood and lymphatic system disorders) | 6 | 2 — Verbatim Terms
Chest Pain or Irregular Heartbeat (Cardiac disorders) | 4 | 6 — Verbatim Terms
Carpal Tunnel (Nervous system disorders) | 0 | 2 — Verbatim Term
Knee Replacement (Surgical and medical procedures) | 0 | 3 — Verbatim Term
Dermatitis, Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 — Verbatim Terms
Rheumatoid Arthritis, Immune Deficiency Syndrome, Multiple Sclerosis, Scleroderma,Autoimmune Disease (Immune system disorders) | 6 | 5 — Verbatim Terms
COPD, Asthma, Emphysema, Chronic Bronchitis, Other Respiratory Problem (Respiratory, thoracic and mediastinal disorders) | 6 | 7 — Verbatim Terms
Sickle Cell Disease (Blood and lymphatic system disorders) | 1 | 0 — Verbatim Term
Legionnaires' Pneumonia (Infections and infestations) | 0 | 1 — Verbatim Terms
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Verbatim Term
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Verbatim Term
Diabetes (Metabolism and nutrition disorders) | 2 | 3 — Verbatim Term
Major Surgery (Surgical and medical procedures) | 6 | 6 — Verbatim Term
Cholesterol, High (Investigations) | 0 | 1
Pituitary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Verbatim Term
COVID-19 (Infections and infestations) | 29 | 29 — Verbatim Term. Not hospitalized
Vertigo (Ear and labyrinth disorders) | 0 | 2
Thyroid Problems (Endocrine disorders) | 0 | 2 — Verbatim Term
Emotional or Psychiatric Problems (Psychiatric disorders) | 3 | 1 — Verbatim Terms
Human Immunodeficiency Virus (HIV) (Immune system disorders) | 1 | 2 — Verbatim Term
Urinary Tract Infections (frequent) (Infections and infestations) | 1 | 0 — Verbatim Term
Broken Toe (Injury, poisoning and procedural complications) | 1 | 0 — Verbatim Term
Pregnant (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Verbatim Term
Ankle, Knee Injury (Injury, poisoning and procedural complications) | 0 | 1 — Verbatim Terms
Perimenopause (possible) (Reproductive system and breast disorders) | 0 | 1 — Verbatim Term
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 — Verbatim Term
Hernia Surgery (Surgical and medical procedures) | 1 | 0 — Verbatim Term
Liver-Related (Hepatobiliary disorders) | 1 | 1 — Fatty liver treated (Usual diet plus Self-Care arm). Fatty liver resolved (Anti-inflammatory dietary intervention arm). Verbatim terms
Concussion (Injury, poisoning and procedural complications) | 1 | 0 — Verbatim Term
Brain Tumor, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Verbatim Term
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0 — Verbatim Term
Bilateral Vein Procedure (Surgical and medical procedures) | 1 | 0 — Verbatim Term. s/p leg cramps
Kidney Stones (Renal and urinary disorders) | 0 | 2 — Verbatim Term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03240406/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03240406/SAP_002.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03240406/ICF_000.pdf